CLINICAL TRIAL: NCT04375280
Title: Evaluation of Impaired Mobility in Chronic Illness Constitution of a Cohort
Acronym: EVALMOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: I-SITE Cap 20-25 project (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2019 COSTES; 2019-A01017-50 (Other: 2019-A01017-50)
Record Dates: First submitted 2020-04-27; First posted 2020-05-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Joint Osteoarthritis; Atherosclerosis of the Distal Arteries, Without Gangrene; Parkinson Disease; Chronic Obstructive Pulmonary Disease, Unspecified; Obesity, Unspecified
Keywords: Prevention; Mobility; Altered mobility; Risk factors; Chronic illness; Chronic pathologies; Physical capacities; Physical test; Activity limitations
MeSH Terms: conditions — Parkinson Disease; Pulmonary Disease, Chronic Obstructive; Obesity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Participants will be involved in a long-term evaluation program combining, body composition measures, physical tests as well as self-administered questionnaires. Participants will be followed for 5 years with evaluations taking place at inclusion, 6 months, at 1, 2 and 5 years
  Interventions: Other: Development of a screening algorithm designed to determine a "dysmobility" profile in patients with chronic illness.

INTERVENTIONS:
Other: Development of a screening algorithm designed to determine a "dysmobility" profile in patients with chronic illness. — Firstly, volunteers will be invited to complete online questionnaires on a secure platform. The mobility assessment will be carried out initially (t1) and up to a maximum of 4 times (t1 to t4) as part of a day hospitalization. Questionnaires will be diverse (SF36, KOOS, HOOS, BROCKER, MNA, TAMPA, etc.) in order to assess several aspects that compose mobility.
  Physical evaluations will include various validated tests (isokinetic strength measure, TUG, 6MWT, Berg Balance Scale, etc.)

SUMMARY:
Chronic illness is a public health issue and mobility loss is frequent in this population. Among its' multiple physical and psychological consequences, increased mortality and cardiovascular morbidity seem the main concern. Therefore, the exploration of locomotor deficiencies, physical capacities and metabolism of patients with chronic illnesses constitutes a major challenge both for the treatment of causal pathologies, as well as for evaluating the impact of therapeutic interventions, the benefit of which will be an improvement in physical capacities and ultimately mobility. In view of the hypothesis of an increase in the prevalence of mobility disorders in this population, this approach is part of a logic of screening and improving the effectiveness of the care of these patients with a multidisciplinary evaluation of individual risks. The EVALMOB protocol was designed in order to try to determine a standard profile of "dysmobility" in patients with chronic illness

DETAILED DESCRIPTION:
We propose to constitute a prospective cohort of subjects carrying chronic disease. The objective is to explore all the different components of mobility (balance, muscle force, body composition, walking ability, metabolism, etc.), to assess their impact on the functional capacity of individuals and to identify their potential interactions. Processing this data could ultimately allow the development of a model to determine a composite standard profile of "dysmobility" in patients with chronic disease.

In the present protocol, parameters will be measured on five occasions (at inclusion, at 6 months from the inclusion day, at 1,2 and 5 year(s) from the inclusion day). All tests will be performed on the same day. New assessments will be done on the same principle as the initial evaluation.

Statistical analyses will be carried out using Stata software (version 13, StataCorp, College Station, USA). Data will be described by frequencies and percentages for categorical variables and by means and standard deviation (or median and interquartile range if data are not normally distributed) for continuous variables. The normality of continuous data will be assessed graphically and using the Shapiro-Wilk test. The main analysis will consist in determining patient profiles regarding their mobility. Clustering-type approaches (supervised or not) will be proposed: k-means, vector machine support, machine learning, factor analysis. For example, factor analyses on mixed data will allow the main components of mobility to be characterized. They can be followed by an ascending hierarchical classification in order to determine homogeneous groups of patients.

These groups will be described and compared on the main criteria evaluated using standard statistical tests: chi2 test (or Fisher's exact test if applicable) for the categorical criteria and using an analysis of variance (or Kruskal-Wallis if data are not normally distributed) for continuous criteria. The main analysis will be broken down more specifically for each of the pathologies considered. In addition, the sensitivity to change will be assessed in each pathology and for each assessment criterion. The search for factors related to the evolution of the different criteria will be carried out using usual tests and mixed multivariate models (logistics for categorical / linear criteria for continuous criteria) considering the subject as a random effect, and adjusting on the time criteria (inclusion / follow-up) and the criteria highlighted in the univariate analyses and in light of the elements reported in the literature. A sensitivity analysis will be proposed in order to study the statistical nature of the missing data and to propose, if necessary, the most suitable method of imputing the data: multiple imputation, maximum bias or LOCF in the case of longitudinal data.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 to 90.
* Patients with chronic pathology contributing to impaired mobility.
* Volunteers who have given their written consent.
* Affiliated to French health care system (for France)

Exclusion Criteria:

* Patients suffering from progressive psychiatric pathologies (active psychosis, hallucinations, etc.) or the presence of another serious unstabilized pathology (decompensated heart failure, progressive terminal cancer, etc.).
* People with poorly controlled or unstable cardiovascular disease.
* Major osteoarticular or neurological problems completely preventing the proper performance of the various tests.
* Non-autonomous patient
* Persons under guardianship, curatorship, deprived of liberty or safeguarding justice.
* People excluded from another study.
* Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2035-08-26 (Estimated); Study Completion 2035-08-26 (Estimated)

PRIMARY OUTCOMES:
dismobility score calculated from the results reported in secondary outcomes | Day 0
  The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles
dismobility score calculated from the results reported in secondary outcomes | Month 6
  The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles
dismobility score calculated from the results reported in secondary outcomes | Year 1
  The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles
dismobility score calculated from the results reported in secondary outcomes | Year 2
  The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles
dismobility score calculated from the results reported in secondary outcomes | Year 5
  The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles

SECONDARY OUTCOMES:
The main objective being to determine patient profiles with regard to "dysmobility", all the criteria detailed as secondary outcomes will be considered for the definition of the profiles | Day 0
  Demographics information will be obtained using a single questionnaire including questions on age, gender, qualification, personal work status, ethnicity, life and occupational events.
Weight (Kg). | Day 0
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Weight (Kg). | Month 6
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Weight (Kg). | Year 1
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Weight (Kg). | Year 2
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Weight (Kg). | Year 5
  Weight will be measured with the medical body weight scale SECA® and according to the ISAK recommendations.
Height (cm). | Day 0
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations
Height (cm). | Month 6
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations
Height (cm). | Year 1
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations
Height (cm). | Year 2
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations
Height (cm). | Year 5
  Height will be measured with a wall mounted tape measure and according to the ISAK recommendations
Body fat percentage (%). | Day 0
  Body fat percentage will be measured with the Harpenden skinfold caliper by measuring skinfold thickness in four different sites (triceps; biceps, suprailiac, subscapular).
Body fat percentage (%). | Month 6
  Body fat percentage will be measured with the Harpenden skinfold caliper by measuring skinfold thickness in four different sites (triceps; biceps, suprailiac, subscapular).
Body fat percentage (%). | Year 1
  Body fat percentage will be measured with the Harpenden skinfold caliper by measuring skinfold thickness in four different sites (triceps; biceps, suprailiac, subscapular).
Body fat percentage (%). | Year 2
  Body fat percentage will be measured with the Harpenden skinfold caliper by measuring skinfold thickness in four different sites (triceps; biceps, suprailiac, subscapular).
Body fat percentage (%). | Year 5
  Body fat percentage will be measured with the Harpenden skinfold caliper by measuring skinfold thickness in four different sites (triceps; biceps, suprailiac, subscapular).
Waist circumference (cm). | Day 0
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Waist circumference (cm). | Month 5
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Waist circumference (cm). | Year 1
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Waist circumference (cm). | Year 2
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Waist circumference (cm). | Year 5
  Waist circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Hip circumference (cm). | Day 0
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm). | Month 6
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm). | Year 1
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm). | Year 2
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Hip circumference (cm). | Year 5
  Hip circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | Day 0
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | Month 6
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | Year 1
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | Year 2
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Brachial circumference (cm). | Year 5
  Brachial circumference will be measured with a medical body tape measure and according to the ISAK recommendations.
Calf circumference (cm). | Day 0
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Calf circumference (cm). | Month 6
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Calf circumference (cm). | Year 1
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Calf circumference (cm). | Year 2
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Calf circumference (cm). | Year 5
  Calf circumference will be measured with a medical body tape measure and according to the ISAK recommendations
Body Mass Index (Kg/m²). | Day 0
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body Mass Index (Kg/m²). | Month 6
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body Mass Index (Kg/m²). | Year 1
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body Mass Index (Kg/m²). | Year 2
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body Mass Index (Kg/m²). | Year 5
  BMI will be calculated (weight in kilograms divided by height in meters squared).
Body composition | Day 0
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Body composition | Month 6
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Body composition | Year 1
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Body composition | Year 2
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
Body composition | Year 5
  Body composition (muscle and fat) will be measured using he Bodystat® Impedance-meter.
T-score (DS). | DAy 0
  - Description: T-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
T-score (DS). | Month 6
  - Description: T-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
T-score (DS). | Year 1
  - Description: T-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
T-score (DS). | Year 2
  - Description: T-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
T-score (DS). | Year 5
  - Description: T-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Z-score (DS). | Day 0
  Z-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Z-score (DS). | Month 6
  Z-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Z-score (DS). | Year 1
  Z-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Z-score (DS). | Year 2
  Z-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Z-score (DS). | Year 5
  Z-score will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Fat mass | Day 0
  Fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mass | Month 6
  Fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mass | Year 1
  Fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mass | Year 2
  Fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mass | Year 5
  Fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass (%). | Day 0
  : Fat free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass (%). | Month 6
  : Fat free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass (%). | Year 1
  : Fat free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass (%). | Year 2
  : Fat free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass (%). | Year 5
  : Fat free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mas index (Kg/m²). | Day 0
  Fat mas index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mas index (Kg/m²). | Month 6
  Fat mas index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mas index (Kg/m²). | Year 1
  Fat mas index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mas index (Kg/m²). | Year 2
  Fat mas index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat mas index (Kg/m²). | Year 5
  Fat mas index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Ratio of android to gynoid fat mass. | Day 0
  Ratio of android to gynoid fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Ratio of android to gynoid fat mass. | Month 6
  Ratio of android to gynoid fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Ratio of android to gynoid fat mass. | Year 1
  Ratio of android to gynoid fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Ratio of android to gynoid fat mass. | Year 2
  Ratio of android to gynoid fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Ratio of android to gynoid fat mass. | Year 5
  Ratio of android to gynoid fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer
Visceral adipose tissue (Kg). | Day 0
  Visceral fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Visceral adipose tissue (Kg). | Month 6
  Visceral fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Visceral adipose tissue (Kg). | Year 1
  Visceral fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Visceral adipose tissue (Kg). | Year 2
  Visceral fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Visceral adipose tissue (Kg). | Year 5
  Visceral fat mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass index (kg/m²). | Day 0
  : Fat-free mass index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass index (kg/m²). | Month 6
  : Fat-free mass index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass index (kg/m²). | Year 1
  : Fat-free mass index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass index (kg/m²). | Year 2
  : Fat-free mass index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Fat-free mass index (kg/m²). | Year 5
  : Fat-free mass index will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Appendicular fat-free mass index (Kg/m²). | Day 0
  Appendicular fat-free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Appendicular fat-free mass index (Kg/m²). | Month 6
  Appendicular fat-free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Appendicular fat-free mass index (Kg/m²). | Year 1
  Appendicular fat-free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Appendicular fat-free mass index (Kg/m²). | Year 2
  Appendicular fat-free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Appendicular fat-free mass index (Kg/m²). | Year 5
  Appendicular fat-free mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Bone mass (Kg) | Day 0
  - Description: Bone mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Bone mass (Kg) | Month 6
  - Description: Bone mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Bone mass (Kg) | Year 1
  - Description: Bone mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Bone mass (Kg) | Year 2
  - Description: Bone mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Bone mass (Kg) | Year 5
  - Description: Bone mass will be measured with the Hologic QDR 4500A dual-energy X-ray absorptiometer.
Daily caloric intake (Kcal/24h). | Day 0
  Daily caloric intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily caloric intake (Kcal/24h). | Month 6
  Daily caloric intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily caloric intake (Kcal/24h). | Year 1
  Daily caloric intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily caloric intake (Kcal/24h). | Year 2
  Daily caloric intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily caloric intake (Kcal/24h). | Year 5
  Daily caloric intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily protein intake (in g and as a percentage of total caloric intake). | Day 0
  Daily protein intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily protein intake (in g and as a percentage of total caloric intake). | Month 6
  Daily protein intake (in g and as a percentage of total caloric intake).
Daily protein intake (in g and as a percentage of total caloric intake). | Year 1
  Daily protein intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily protein intake (in g and as a percentage of total caloric intake). | Year 2
  Daily protein intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily protein intake (in g and as a percentage of total caloric intake). | Year 5
  Daily protein intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily carbohydrate intake (in g and as a percentage of total caloric intake). | Day 0
  Daily carbohydrate intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily carbohydrate intake (in g and as a percentage of total caloric intake). | Month 6
  Daily carbohydrate intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily carbohydrate intake (in g and as a percentage of total caloric intake). | Year 1
  Daily carbohydrate intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily carbohydrate intake (in g and as a percentage of total caloric intake). | Year 2
  Daily carbohydrate intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily carbohydrate intake (in g and as a percentage of total caloric intake). | Year 5
  Daily carbohydrate intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily fat intake (in g and as a percentage of total caloric intake). | Day 0
  Daily fat intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily fat intake (in g and as a percentage of total caloric intake). | Month 6
  Daily fat intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily fat intake (in g and as a percentage of total caloric intake). | Year 1
  Daily fat intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily fat intake (in g and as a percentage of total caloric intake). | Year 2
  Daily fat intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Daily fat intake (in g and as a percentage of total caloric intake). | Year 5
  Daily fat intake will be estimated with a 24-hour (all foods and beverages consumed by the respondent in the past 24 hours).
Nutritional status assessment | Day 0
  Nutritional status assessment will be assessed with the Mini Nutritional Assessment Questionnaire.
Nutritional status assessment | Month 6
  Nutritional status assessment will be assessed with the Mini Nutritional Assessment Questionnaire.
Nutritional status assessment | Year 1
  Nutritional status assessment will be assessed with the Mini Nutritional Assessment Questionnaire.
Nutritional status assessment | Year 2
  Nutritional status assessment will be assessed with the Mini Nutritional Assessment Questionnaire.
Nutritional status assessment | Year 5
  Nutritional status assessment will be assessed with the Mini Nutritional Assessment Questionnaire.
Risk of undernutrition. | Day 0
  Risk of undernutrition will be assessed with the Brocker Questionnaire
Risk of undernutrition. | Month 6
  Risk of undernutrition will be assessed with the Brocker Questionnaire
Risk of undernutrition. | Year 1
  Risk of undernutrition will be assessed with the Brocker Questionnaire
Risk of undernutrition. | Year 2
  Risk of undernutrition will be assessed with the Brocker Questionnaire
Risk of undernutrition. | Year 5
  Risk of undernutrition will be assessed with the Brocker Questionnaire
Basic biology. | Day 0
  : Basic biology will be measured using endocrine assays (fasting blood glucose, HbA1c, HDL-c and LDL-c, TG, CPK)
Basic biology. | Month 6
  : Basic biology will be measured using endocrine assays (fasting blood glucose, HbA1c, HDL-c and LDL-c, TG, CPK)
Basic biology. | Year 1
  : Basic biology will be measured using endocrine assays (fasting blood glucose, HbA1c, HDL-c and LDL-c, TG, CPK)
Basic biology. | Year 2
  : Basic biology will be measured using endocrine assays (fasting blood glucose, HbA1c, HDL-c and LDL-c, TG, CPK)
Basic biology. | Year 5
  : Basic biology will be measured using endocrine assays (fasting blood glucose, HbA1c, HDL-c and LDL-c, TG, CPK)
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Day 0
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Month 6
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Year 1
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Year 2
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isometric strength of the quadriceps muscles at 45° (Nm). | Year 5
  : Maximum voluntary isometric strength of the quadriceps muscles will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Day 0
  - Description: Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Month 6
  - Description: Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Year 1
  - Description: Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Year 2
  - Description: Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s (Nm). | Year 5
  - Description: Maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Month 6
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Year 1
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Year 2
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s (Nm). | Year 5
  Maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Day 0
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Month 6
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Year 1
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Year 2
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s (eccentric contraction) (Nm). | Year 5
  Maximum voluntary isokinetic strength of the quadriceps muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Day 0
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Month 6
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Year 1
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Year 2
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s (Nm). | Year 5
  Maximum voluntary isokinetic strength of the hamstring muscles at 60°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Day 0
  - Description: Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Month 6
  - Description: Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Year 1
  - Description: Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Year 2
  - Description: Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s (Nm). | Year 5
  - Description: Maximum voluntary isokinetic strength of the hamstring muscles at 240°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Day 0
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Month 6
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Year 1
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Year 2
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) (Nm). | Year 5
  Maximum voluntary isokinetic strength of the hamstring muscles at 30°/s will be measured with the HUMA® /NORM™ device.
Endurance coefficient of the quadriceps muscles at 180°/s. | Day 0
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device.
Endurance coefficient of the quadriceps muscles at 180°/s. | Month 6
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device.
Endurance coefficient of the quadriceps muscles at 180°/s. | Year 1
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device.
Endurance coefficient of the quadriceps muscles at 180°/s. | Year 2
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device.
Endurance coefficient of the quadriceps muscles at 180°/s. | Year 5
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device.
Endurance coefficient of the hamstring muscles at 180°/s. | Day 0
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device..
Endurance coefficient of the hamstring muscles at 180°/s. | Month 6
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device..
Endurance coefficient of the hamstring muscles at 180°/s. | Year 1
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device..
Endurance coefficient of the hamstring muscles at 180°/s. | Year 2
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device..
Endurance coefficient of the hamstring muscles at 180°/s. | Year 5
  Endurance coefficient will be estimated as a Σ Peak torque ratio of the last 3 contractions on the first 3 at 180°/s with the HUMA® /NORM™ device..
Functional ratio | Day 0
  Functional ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 60°/s with the maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s.
Functional ratio | Month 6
  Functional ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 60°/s with the maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s.
Functional ratio | Year 1
  Functional ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 60°/s with the maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s.
Functional ratio | Year 2
  Functional ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 60°/s with the maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s.
Functional ratio | Year 5
  Functional ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 60°/s with the maximum voluntary isokinetic strength of the quadriceps muscles at 60°/s.
Mixed ratio | Day 0
  - Mixed ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) with the maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s Title: Maximum voluntary strength of the quadriceps muscles at 60°/s.
Mixed ratio | Month 6
  - Mixed ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) with the maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s Title: Maximum voluntary strength of the quadriceps muscles at 60°/s.
Mixed ratio | Year 1
  - Mixed ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) with the maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s Title: Maximum voluntary strength of the quadriceps muscles at 60°/s.
Mixed ratio | Year 2
  - Mixed ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) with the maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s Title: Maximum voluntary strength of the quadriceps muscles at 60°/s.
Mixed ratio | Year 5
  - Mixed ratio will be estimated by dividing the maximum voluntary isokinetic strength of the hamstring muscles at 30°/s (eccentric contraction) with the maximum voluntary isokinetic strength of the quadriceps muscles at 240°/s Title: Maximum voluntary strength of the quadriceps muscles at 60°/s.
Maximum voluntary hand grip strength (Kg). | Day 0
  Maximum voluntary hand grip strength will be measured with the Jamar® hydraulic dynamometer and with the Baseline® pneumatic dynamometer.
Maximum voluntary hand grip strength (Kg). | Month 6
  Maximum voluntary hand grip strength will be measured with the Jamar® hydraulic dynamometer and with the Baseline® pneumatic dynamometer.
Maximum voluntary hand grip strength (Kg). | Year 1
  Maximum voluntary hand grip strength will be measured with the Jamar® hydraulic dynamometer and with the Baseline® pneumatic dynamometer.
Maximum voluntary hand grip strength (Kg). | Year 2
  Maximum voluntary hand grip strength will be measured with the Jamar® hydraulic dynamometer and with the Baseline® pneumatic dynamometer.
Maximum voluntary hand grip strength (Kg). | Year 5
  Maximum voluntary hand grip strength will be measured with the Jamar® hydraulic dynamometer and with the Baseline® pneumatic dynamometer.
Maximum voluntary pinch strength (Kg). | Day 0
  Maximum voluntary pinch strength will be measured with the Baseline® pinch gauche test mechanical dynamometer.
Maximum voluntary pinch strength (Kg). | Month 6
  Maximum voluntary pinch strength will be measured with the Baseline® pinch gauche test mechanical dynamometer.
Maximum voluntary pinch strength (Kg). | Year 1
  Maximum voluntary pinch strength will be measured with the Baseline® pinch gauche test mechanical dynamometer.
Maximum voluntary pinch strength (Kg). | Year 2
  Maximum voluntary pinch strength will be measured with the Baseline® pinch gauche test mechanical dynamometer.
Maximum voluntary pinch strength (Kg). | Year 5
  Maximum voluntary pinch strength will be measured with the Baseline® pinch gauche test mechanical dynamometer.
Hip passive joint range | Day 0
  Hip joint range will be measured with a medical goniometer.
Hip passive joint range | Month 6
  Hip joint range will be measured with a medical goniometer.
Hip passive joint range | Year 1
  Hip joint range will be measured with a medical goniometer.
Hip passive joint range | Year 2
  Hip joint range will be measured with a medical goniometer.
Hip passive joint range | Year 5
  Hip joint range will be measured with a medical goniometer.
Knee passive joint range. | Day 0
  Knee joint range will be measured with a medical goniometer.
Knee passive joint range. | Month 6
  Knee joint range will be measured with a medical goniometer.
Knee passive joint range. | Year 1
  Knee joint range will be measured with a medical goniometer.
Knee passive joint range. | Year 2
  Knee joint range will be measured with a medical goniometer.
Knee passive joint range. | Year 5
  Knee joint range will be measured with a medical goniometer.
Ankle passive joint range | Day 0
  Ankle joint range will be measured with a medical goniometer.
Ankle passive joint range | Month 6
  Ankle joint range will be measured with a medical goniometer.
Ankle passive joint range | Year 1
  Ankle joint range will be measured with a medical goniometer.
Ankle passive joint range | Year 2
  Ankle joint range will be measured with a medical goniometer.
Ankle passive joint range | Year 5
  Ankle joint range will be measured with a medical goniometer.
Lower and upper limb muscle power assessment (MRC) | Day 0
  Lower and upper limb muscle power assessment will be performed by an experienced physician.
Lower and upper limb muscle power assessment (MRC) | Month 6
  Lower and upper limb muscle power assessment will be performed by an experienced physician.
Lower and upper limb muscle power assessment (MRC) | Year 1
  Lower and upper limb muscle power assessment will be performed by an experienced physician.
Lower and upper limb muscle power assessment (MRC) | Year 2
  Lower and upper limb muscle power assessment will be performed by an experienced physician.
Lower and upper limb muscle power assessment (MRC) | Year 5
  Lower and upper limb muscle power assessment will be performed by an experienced physician.
Statokinesigram surface area (mm²) | Day 0
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Statokinesigram surface area (mm²) | Month 6
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Statokinesigram surface area (mm²) | Year 1
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Statokinesigram surface area (mm²) | Year 2
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Statokinesigram surface area (mm²) | Year 5
  Statokinesigram surface area will be measured with the STATIPRO® static posturography platform.
Stabilogram length (mm). | Day 0
  Stabilogram length will be measured with the STATIPRO® static posturography platform
Stabilogram length (mm). | Month 6
  Stabilogram length will be measured with the STATIPRO® static posturography platform
Stabilogram length (mm). | Year 1
  Stabilogram length will be measured with the STATIPRO® static posturography platform
Stabilogram length (mm). | Year 2
  Stabilogram length will be measured with the STATIPRO® static posturography platform
Stabilogram length (mm). | Year 5
  Stabilogram length will be measured with the STATIPRO® static posturography platform
Maximal deflection (forward, backward left and right). | Day 0
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Maximal deflection (forward, backward left and right). | Month 6
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Maximal deflection (forward, backward left and right). | Year 1
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Maximal deflection (forward, backward left and right). | Year 2
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Maximal deflection (forward, backward left and right). | Year 5
  Maximal deflection will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Day 0
  : Velocity variations will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Month 6
  : Velocity variations will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Year 1
  : Velocity variations will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Year 2
  : Velocity variations will be measured with the STATIPRO® static posturography platform.
Velocity variations (mm/s). | Year 5
  : Velocity variations will be measured with the STATIPRO® static posturography platform.
: Romberg ratio according to sway area | Day 0
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
: Romberg ratio according to sway area | Month 6
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
: Romberg ratio according to sway area | Year 1
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
: Romberg ratio according to sway area | Year 2
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
: Romberg ratio according to sway area | Year 5
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to center of pressure path length | Day 0
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to center of pressure path length | Month 6
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to center of pressure path length | Year 1
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to center of pressure path length | Year 2
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
Romberg ratio according to center of pressure path length | Year 5
  Romberg ratio will be measured with the STATIPRO® static posturography platform.
: Plantar pressure ratio sway area. | Day 0
  Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform.
: Plantar pressure ratio sway area. | Month 6
  Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform.
: Plantar pressure ratio sway area. | Year 1
  Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform.
: Plantar pressure ratio sway area. | Year 2
  Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform.
: Plantar pressure ratio sway area. | Year 5
  Plantar pressure ratio sway area will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio length. | Day 0
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio length. | Month 6
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio length. | Year 1
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio length. | Year 2
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Plantar pressure ratio length. | Year 5
  Plantar pressure ratio length will be measured with the STATIPRO® static posturography platform.
Walking velocity (cm/s). | Day 0
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Walking velocity (cm/s). | Month 6
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Walking velocity (cm/s). | Year 1
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Walking velocity (cm/s). | Year 2
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Walking velocity (cm/s). | Year 5
  Walking velocity will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | Day 0
  : Cadence will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | Month 6
  : Cadence will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | Year 1
  : Cadence will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | Year 2
  : Cadence will be measured with the GAITRite® Electronic Walkway.
Cadence (steps/min). | Year 5
  : Cadence will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | DAy 0
  Step length will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | Month 6
  Step length will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | Year 1
  Step length will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | Year 2
  Step length will be measured with the GAITRite® Electronic Walkway.
Step length (left and right foot) (cm) | Year 5
  Step length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | Day 0
  Stride length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | month 6
  Stride length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | year 1
  Stride length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | year 2
  Stride length will be measured with the GAITRite® Electronic Walkway.
Stride length (cm). | year 5
  Stride length will be measured with the GAITRite® Electronic Walkway.
Single support time left and right foot (s). | Day 0
  Single support time will be measured with the GAITRite® Electronic Walkway.
Single support time left and right foot (s). | Month 6
  Single support time will be measured with the GAITRite® Electronic Walkway.
Single support time left and right foot (s). | Year 1
  Single support time will be measured with the GAITRite® Electronic Walkway.
Single support time left and right foot (s). | Year 2
  Single support time will be measured with the GAITRite® Electronic Walkway.
Single support time left and right foot (s). | Year 5
  Single support time will be measured with the GAITRite® Electronic Walkway.
Double support time (s). | Day 0
  : Double support time will be measured with the GAITRite® Electronic Walkway.
Double support time (s). | Month 6
  : Double support time will be measured with the GAITRite® Electronic Walkway.
Double support time (s). | YEar 1
  : Double support time will be measured with the GAITRite® Electronic Walkway.
Double support time (s). | Year 2
  : Double support time will be measured with the GAITRite® Electronic Walkway.
Double support time (s). | Year 5
  : Double support time will be measured with the GAITRite® Electronic Walkway.
Swing time (s). | Day 0
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing time (s). | Month 6
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing time (s). | Year 1
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing time (s). | Year 2
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing time (s). | Year 5
  : Swing time will be measured with the GAITRite® Electronic Walkway.
Swing phase (as a % of walking cycle). | DAy 0
  : Swing phase will be measured with the GAITRite® Electronic Walkway.
Swing phase (as a % of walking cycle). | Month 6
  : Swing phase will be measured with the GAITRite® Electronic Walkway.
Swing phase (as a % of walking cycle). | Year 1
  : Swing phase will be measured with the GAITRite® Electronic Walkway.
Swing phase (as a % of walking cycle). | Year 2
  : Swing phase will be measured with the GAITRite® Electronic Walkway.
Swing phase (as a % of walking cycle). | Year 5
  : Swing phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (as a % of walking cycle). | Day 0
  Stance phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (as a % of walking cycle). | Month 6
  Stance phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (as a % of walking cycle). | Year 1
  Stance phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (as a % of walking cycle). | Year 2
  Stance phase will be measured with the GAITRite® Electronic Walkway.
Stance phase (as a % of walking cycle). | Year 5
  Stance phase will be measured with the GAITRite® Electronic Walkway.
Vo2max (maximal oxygen consumption) (mL/Kg/min). | Day 0
  : Vo2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Vo2max (maximal oxygen consumption) (mL/Kg/min). | Month 6
  : Vo2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Vo2max (maximal oxygen consumption) (mL/Kg/min). | Year 1
  : Vo2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Vo2max (maximal oxygen consumption) (mL/Kg/min). | Year 2
  : Vo2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Vo2max (maximal oxygen consumption) (mL/Kg/min). | Year 5
  : Vo2max will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum heart rate (bpm). | Day 0
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum heart rate (bpm). | Month 6
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum heart rate (bpm). | Year 1
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum heart rate (bpm). | Year 2
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum heart rate (bpm). | Year 5
  Maximum heart rate will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts). | Day 0
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts). | Month 6
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts). | Year 1
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts). | Year 2
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Maximum power (Watts). | Year 5
  Maximum power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold power (Watts). | Day 0
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold power (Watts). | Month 6
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold power (Watts). | Year 1
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold power (Watts). | Year 2
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold power (Watts). | Year 5
  Threshold power will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold heart rate (bpm). | DAy 0
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold heart rate (bpm). | Month 6
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold heart rate (bpm). | Year 1
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold heart rate (bpm). | Year 2
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Threshold heart rate (bpm). | Year 5
  Threshold heart will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Forced vital Capacity (L). | Day 0
  : Forced vital Capacity will be measured with a spirometry test.
Forced vital Capacity (L). | Month 6
  : Forced vital Capacity will be measured with a spirometry test.
Forced vital Capacity (L). | Year 1
  : Forced vital Capacity will be measured with a spirometry test.
Forced vital Capacity (L). | Year 2
  : Forced vital Capacity will be measured with a spirometry test.
Forced vital Capacity (L). | Year 5
  : Forced vital Capacity will be measured with a spirometry test.
Forced Expiratory volume (L) | Day 0
  Forced Expiratory volume will be measured with a spirometry test.
Forced Expiratory volume (L) | Month 6
  Forced Expiratory volume will be measured with a spirometry test.
Forced Expiratory volume (L) | Year 1
  Forced Expiratory volume will be measured with a spirometry test.
Forced Expiratory volume (L) | Year 2
  Forced Expiratory volume will be measured with a spirometry test.
Forced Expiratory volume (L) | Year 5
  Forced Expiratory volume will be measured with a spirometry test.
Tiffeneau ratio (%). | Day 0
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Tiffeneau ratio (%). | Month 6
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Tiffeneau ratio (%). | Year 1
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Tiffeneau ratio (%). | Year 2
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Tiffeneau ratio (%). | Year 5
  Tiffeneau ratio will be calculated by dividing the Forced Expiratory volume to the Forced vital Capacity.
Ventilatory reserve (%). | Day 0
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Ventilatory reserve (%). | Month 6
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Ventilatory reserve (%). | Year 1
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Ventilatory reserve (%). | Year 2
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Ventilatory reserve (%). | Year 5
  Ventilatory reserve will be obtained by performing a cardiopulmonary exercise testing at maximal effort during incremental exercise on a cycle ergometer.
Physical activity | Day 0
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Physical activity | Month 6
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Physical activity | Year 1
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Physical activity | Year 2
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Physical activity | Year 5
  Physical activity will be measured using the Global Physical Activity Questionnaire (GPAQ)
Functional capacity timed-up and go | Day 0
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity timed-up and go | Month 6
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity timed-up and go | Year 1
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity timed-up and go | Year 2
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity timed-up and go | Year 5
  Functional capacity will be evaluated using the Timed-Up and Go test.
Functional capacity TDM6 | Day 0
  Functional capacity will be evaluated using the 6-minute walk test.
Functional capacity TDM6 | Month 6
  Functional capacity will be evaluated using the 6-minute walk test.
Functional capacity TDM6 | Year 1
  Functional capacity will be evaluated using the 6-minute walk test.
Functional capacity TDM6 | Year 2
  Functional capacity will be evaluated using the 6-minute walk test.
Functional capacity TDM6 | Year 5
  Functional capacity will be evaluated using the 6-minute walk test.
Functional capacity Five Times Sit to Stand test. | Day 0
  Functional capacity will be evaluated using the Five Times Sit to Stand test.
Functional capacity Five Times Sit to Stand test. | Month 6
  Functional capacity will be evaluated using the Five Times Sit to Stand test.
Functional capacity Five Times Sit to Stand test. | Year 1
  Functional capacity will be evaluated using the Five Times Sit to Stand test.
Functional capacity Five Times Sit to Stand test. | Year 2
  Functional capacity will be evaluated using the Five Times Sit to Stand test.
Functional capacity Five Times Sit to Stand test. | Year 5
  Functional capacity will be evaluated using the Five Times Sit to Stand test.
Functional capacity SPPB | Day 0
  Functional capacity will be evaluated using the Five Times Sit to Stand test.Functional capacity will be evaluated using the Short Physical Performance Battery test.
Functional capacity SPPB | Month 6
  Functional capacity will be evaluated using the Five Times Sit to Stand test.Functional capacity will be evaluated using the Short Physical Performance Battery test.
Functional capacity SPPB | Year 1
  Functional capacity will be evaluated using the Five Times Sit to Stand test.Functional capacity will be evaluated using the Short Physical Performance Battery test.
Functional capacity SPPB | Year 2
  Functional capacity will be evaluated using the Five Times Sit to Stand test.Functional capacity will be evaluated using the Short Physical Performance Battery test.
Functional capacity SPPB | Year 5
  Functional capacity will be evaluated using the Five Times Sit to Stand test.Functional capacity will be evaluated using the Short Physical Performance Battery test.
Functional capacity the mini-BESTest. | Day 0
  Functional capacity will be evaluated using the mini-BESTest.
Functional capacity the mini-BESTest. | Month 6
  Functional capacity will be evaluated using the mini-BESTest.
Functional capacity the mini-BESTest. | Year 1
  Functional capacity will be evaluated using the mini-BESTest.
Functional capacity the mini-BESTest. | Year 2
  Functional capacity will be evaluated using the mini-BESTest.
Functional capacity the mini-BESTest. | Year 5
  Functional capacity will be evaluated using the mini-BESTest.
Functional capacity Berg Balance Scale. | Day 0
  Functional capacity will be evaluated using the Berg Balance Scale.
Functional capacity Berg Balance Scale. | Month 6
  Functional capacity will be evaluated using the Berg Balance Scale.
Functional capacity Berg Balance Scale. | Year 1
  Functional capacity will be evaluated using the Berg Balance Scale.
Functional capacity Berg Balance Scale. | Year 2
  Functional capacity will be evaluated using the Berg Balance Scale.
Functional capacity Berg Balance Scale. | Year 5
  Functional capacity will be evaluated using the Berg Balance Scale.
Functional capacity 10-meter walk test | Day 0
  Functional capacity will be evaluated using the 10-meter walk test (at usual and maximal pace).
Functional capacity 10-meter walk test | Month 6
  Functional capacity will be evaluated using the 10-meter walk test (at usual and maximal pace).
Functional capacity 10-meter walk test | Year 1
  Functional capacity will be evaluated using the 10-meter walk test (at usual and maximal pace).
Functional capacity 10-meter walk test | Year 2
  Functional capacity will be evaluated using the 10-meter walk test (at usual and maximal pace).
Functional capacity 10-meter walk test | Year 5
  Functional capacity will be evaluated using the 10-meter walk test (at usual and maximal pace).
Dyspnea | Day 0
  Dyspnea will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Dyspnea | Month 6
  Dyspnea will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Dyspnea | Year 1
  Dyspnea will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Dyspnea | Year 2
  Dyspnea will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Dyspnea | Year 5
  Dyspnea will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Perceived exertion before, during and after effort | DAy 0
  Perceived exertion will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Perceived exertion before, during and after effort | Month 6
  Perceived exertion will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Perceived exertion before, during and after effort | Year 1
  Perceived exertion will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Perceived exertion before, during and after effort | Year 2
  Perceived exertion will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Perceived exertion before, during and after effort | Year 5
  Perceived exertion will be evaluated by a Numeric Rating scale ranging from 0 to 10.
Pain | Day 0
  : Pain will be measured by a visual analogue scale (VAS) ranging from 0 to 10 and possibly as appropriate by other questionnaires or specific scales.
Pain | Month 6
  : Pain will be measured by a visual analogue scale (VAS) ranging from 0 to 10 and possibly as appropriate by other questionnaires or specific scales.
Pain | Year 1
  : Pain will be measured by a visual analogue scale (VAS) ranging from 0 to 10 and possibly as appropriate by other questionnaires or specific scales.
Pain | Year 2
  : Pain will be measured by a visual analogue scale (VAS) ranging from 0 to 10 and possibly as appropriate by other questionnaires or specific scales.
Pain | Year 5
  : Pain will be measured by a visual analogue scale (VAS) ranging from 0 to 10 and possibly as appropriate by other questionnaires or specific scales.
Sarcopenia risk | Day 0
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Sarcopenia risk | Month 6
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Sarcopenia risk | Year 1
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Sarcopenia risk | Year 2
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Sarcopenia risk | Year 5
  Sarcopenia risk will be evaluated with the SARC-F Questionnaire.
Social insecurity | Day 0
  Social insecurity will be evaluated with the EPICES Score Questionnaire.
Social insecurity | Month 6
  Social insecurity will be evaluated with the EPICES Score Questionnaire.
Social insecurity | Year 1
  Social insecurity will be evaluated with the EPICES Score Questionnaire.
Social insecurity | Year 2
  Social insecurity will be evaluated with the EPICES Score Questionnaire.
Social insecurity | Year 5
  Social insecurity will be evaluated with the EPICES Score Questionnaire.
Kinesiophobia | Day 0
  Kinesiophobia will be evaluated with the TAMPA Scale.
Kinesiophobia | Month 6
  Kinesiophobia will be evaluated with the TAMPA Scale.
Kinesiophobia | Year 1
  Kinesiophobia will be evaluated with the TAMPA Scale.
Kinesiophobia | Year 2
  Kinesiophobia will be evaluated with the TAMPA Scale.
Kinesiophobia | Year 5
  Kinesiophobia will be evaluated with the TAMPA Scale.
Quality of life | Day 0
  Quality of life will be evaluated with the 36-Item Short Form Survey.
Quality of life | Month 6
  Quality of life will be evaluated with the 36-Item Short Form Survey.
Quality of life | Year 1
  Quality of life will be evaluated with the 36-Item Short Form Survey.
Quality of life | Year 2
  Quality of life will be evaluated with the 36-Item Short Form Survey.
Quality of life | Year 5
  Quality of life will be evaluated with the 36-Item Short Form Survey.
: Balance confidence in performing various activities | Day 0
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.vey.
: Balance confidence in performing various activities | Month 6
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.vey.
: Balance confidence in performing various activities | Year 1
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.vey.
: Balance confidence in performing various activities | Year 2
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.vey.
: Balance confidence in performing various activities | Year 5
  Self-report balance confidence will be evaluated with the Activities-specific Balance Confidence (ABC) Scale.vey.
Functioning in regards to activities of daily living. | Day 0
  Functioning will be evaluated with the Lawton Instrumental Activities of Daily Living (IADL) Scale.
Functioning in regards to activities of daily living. | Month 6
  Functioning will be evaluated with the Lawton Instrumental Activities of Daily Living (IADL) Scale.
Functioning in regards to activities of daily living. | Year 1
  Functioning will be evaluated with the Lawton Instrumental Activities of Daily Living (IADL) Scale.
Functioning in regards to activities of daily living. | Year 2
  Functioning will be evaluated with the Lawton Instrumental Activities of Daily Living (IADL) Scale.
Functioning in regards to activities of daily living. | Year 5
  Functioning will be evaluated with the Lawton Instrumental Activities of Daily Living (IADL) Scale.
Exhaustion | Day 0
  Exhaustion will be evaluated with the FACIT-F Questionnaire.
Exhaustion | Month 6
  Exhaustion will be evaluated with the FACIT-F Questionnaire.
Exhaustion | Year 1
  Exhaustion will be evaluated with the FACIT-F Questionnaire.
Exhaustion | Year 2
  Exhaustion will be evaluated with the FACIT-F Questionnaire.
Exhaustion | Year 5
  Exhaustion will be evaluated with the FACIT-F Questionnaire.
Patient's opinion about their knee and associated problems | Day 0
  : Outcomes will be evaluated with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Patient's opinion about their knee and associated problems | Month 6
  : Outcomes will be evaluated with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Patient's opinion about their knee and associated problems | Year 1
  : Outcomes will be evaluated with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Patient's opinion about their knee and associated problems | Year 2
  : Outcomes will be evaluated with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Patient's opinion about their knee and associated problems | Year 5
  : Outcomes will be evaluated with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Patient's opinion about their hip and associated problems | Day 0
  Outcomes will be evaluated with the Hip Injury and Osteoarthritis Outcome Score (HOOS).
Patient's opinion about their hip and associated problems | Month 6
  Outcomes will be evaluated with the Hip Injury and Osteoarthritis Outcome Score (HOOS).
Patient's opinion about their hip and associated problems | Year 1
  Outcomes will be evaluated with the Hip Injury and Osteoarthritis Outcome Score (HOOS).
Patient's opinion about their hip and associated problems | Year 2
  Outcomes will be evaluated with the Hip Injury and Osteoarthritis Outcome Score (HOOS).
Patient's opinion about their hip and associated problems | Year 5
  Outcomes will be evaluated with the Hip Injury and Osteoarthritis Outcome Score (HOOS).
Predicting discharge destination after total joint arthroplasty. | Day 0
  : Discharge destination will be evaluated with the Risk Assessment and Prediction Tool (RAPT);
Predicting discharge destination after total joint arthroplasty. | Month 6
  : Discharge destination will be evaluated with the Risk Assessment and Prediction Tool (RAPT);
Physical function in myositis patients | Day 0
  Physical function will be evaluated with the Stanford Health Assessment Questionnaire.
Physical function in myositis patients | Month 6
  Physical function will be evaluated with the Stanford Health Assessment Questionnaire.
Physical function in myositis patients | Year 1
  Physical function will be evaluated with the Stanford Health Assessment Questionnaire.
Physical function in myositis patients | Year 2
  Physical function will be evaluated with the Stanford Health Assessment Questionnaire.
Physical function in myositis patients | Year 5
  Physical function will be evaluated with the Stanford Health Assessment Questionnaire.
Quality of life in Parkinson's Disease | Day 0
  Quality of life will be measured with the Parkinson's Disease Questionnaire-39 (PDQ-39).
Quality of life in Parkinson's Disease | Month 6
  Quality of life will be measured with the Parkinson's Disease Questionnaire-39 (PDQ-39).
Quality of life in Parkinson's Disease | Year 1
  Quality of life will be measured with the Parkinson's Disease Questionnaire-39 (PDQ-39).
Quality of life in Parkinson's Disease | Year 2
  Quality of life will be measured with the Parkinson's Disease Questionnaire-39 (PDQ-39).
Quality of life in Parkinson's Disease | Year 5
  Quality of life will be measured with the Parkinson's Disease Questionnaire-39 (PDQ-39).
Actimetry. | during 5 consecutive days after day 0
  Actimetry data (energy expenditure, number of steps, sedentary time, total physical activity, etc.) will be obtained with the WGT3X-BT Actigraph inertial sensor unit.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Costes, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France